CLINICAL TRIAL: NCT02235870
Title: The Six-Month Adjunctive Weight Reduction Therapy (SMART) Trial
Brief Title: Obalon Balloon System Pivotal IDE (SMART) Trial
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obalon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTL-1100-0013
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Weight Loss; Obesity; BMI
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): In accordance with the randomization assignment, treatment arm subjects will receive a 6-month course of Balloon therapy with a nutrition and lifestyle program. Balloon treatment consists of placement of 3 balloons Obalon Intragastric Balloons in the first 3 months of therapy.
  Interventions: Device: Obalon Intragastric Balloons; Behavioral: Nutrition and Lifestyle Program
- Control Group (Sham Comparator): Control arm subjects will receive a single 6-month course of sham device therapy with a nutrition and lifestyle program. Sham treatment consists of placement of 3 shams in the first 3 months of therapy.
  Interventions: Device: Sham Device; Behavioral: Nutrition and Lifestyle Program

INTERVENTIONS:
Device: Obalon Intragastric Balloons — Intragastric Balloon System to aid in portion control.
  Arms: Treatment Group
Device: Sham Device — Sham Intragastric Balloon
  Arms: Control Group
Behavioral: Nutrition and Lifestyle Program — Nutrition and lifestyle program reviewed with subjects every 3 weeks for 6 months.

SUMMARY:
This pivotal trial of the Obalon Balloon System is intended to generate safety and effectiveness data required to support a future marketing application. The trial has been designed to evaluate a 6-month use of the Obalon Balloon System as an adjunct to a nutrition and lifestyle behavior modification program.

Weight loss will be evaluated after the 6-month course to determine if a specific predefined superiority margin can be achieved in the device group compared to a sham-control group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 22-64 years
2. Current BMI of 30.0 - 40 kg/m2
3. Previously attempted to lose weight unsuccessfully using a medically supervised or non-medically supervised diet
4. Willing to attend all protocol-specified follow-up visits plus any additional follow-up visits as required throughout the entire study period
5. Willing to avoid non-commercial air travel and scuba diving during the entire study period
6. Willing to avoid medications or other substances known to effect weight changes during the study
7. Willing to avoid Non-Steroidal Anti-inflammatory Drugs (NSAIDs) or other medications known to be gastric irritants during the study
8. Willing to use contraception and avoid pregnancy during the study if the subject is female with child bearing potential
9. Willing to provide written informed consent

Exclusion Criteria:

1. Significant weight loss in the past 12 months
2. Use of medications or other substances known to induce weight gain or weight loss
3. Participation in any clinical study at the start of this trial or in the last year
4. Known history of endocrine disorders affecting weight
5. Currently receiving chronic steroid or immunosuppressive therapy or has previously been diagnosed with HIV
6. Subjects diagnosed with bulimia, binge eating, compulsive overeating, high liquid calorie intake habits or similar eating related psychological disorders
7. Intent to undergo gastric surgery or gastric banding during the study period or within the 6 month period after completion of this study
8. Prior use of any weight loss medical device
9. Known history of structural or functional disorders of the esophagus
10. Known history of structural or functional disorder of the esophagus, including any swallowing disorder, esophageal chest pain disorders, or drug refractory esophageal reflux symptoms
11. Known history of structural or functional disorders of the stomach
12. Known history of a structural or functional disorder of the stomach, including any symptoms of chronic upper abdominal pain, chronic nausea, chronic vomiting, chronic dyspepsia or symptoms suggestive of gastroparesis, including post-prandial fullness or pain, post-prandial nausea or vomiting or early satiety
13. Known history of duodenal ulcer, intestinal diverticula (diverticulitis), intestinal varices, intestinal stricture/stenosis, small bowel obstruction, or any other obstructive disorder of the gastrointestinal (GI) tract
14. Currently have ongoing symptoms suggestive of intermittent small bowel obstruction, such as recurrent bouts of post-prandial abdominal pain, nausea or vomiting
15. Known history irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease
16. Known history of GI surgeries that may have resulted in anatomical GI tract abnormalities
17. Type 1 diabetes
18. Type 2 diabetes requiring insulin or other hypoglycemic oral agents.
19. Experienced a myocardial infarction, has a known history of angina, a known history of congestive heart failure, or is currently being medically treated for any other cardiac condition
20. Poorly controlled hypertension, (≥ 160 mmHg Systolic and ≥ 100mmHg Diastolic).
21. End stage renal disease or requiring hemodialysis within the past 6 months
22. Unwilling or unable to avoid Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), including Aspirin, Diclofenac, Ibuprofen, Naproxen, or other medications known to be gastric irritants beginning two weeks prior to enrollment and throughout the entire study period
23. Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying
24. Subjects requiring the use of anti-platelet drugs or other agents affecting the normal clotting of blood
25. Untreated or unstable alcohol or illicit drug addiction
26. Known history of allergies to any component of the device materials
27. Currently pregnant or breastfeeding or intention of becoming pregnant during the study
28. Life expectancy less than 1 year or severe renal, hepatic, pulmonary or other medical condition, in the opinion of the investigator
29. Subject is employed by the investigator, or is a close relative of the investigator, or the investigator's staff
30. Subject is a close relative of another subject already enrolled in the study.
31. Any other condition that, in the opinion of the investigator, would interfere with subject participation, may confound the study results, or interfere with compliance with the study (e.g., psychosocial issues).

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 711 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy VandenBerg, Study Chair — Obalon Therapeutics, Inc.
Locations (15):
- United States (15):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Southern California Research Center, Coronado, California
  - Bariatric Institute of Greater Chicago, Hinsdale, Illinois
  - Endoscopic Microsurgery Associates, Towson, Maryland
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University Hospital in St. Louis, St Louis, Missouri
  - Stony Brook Medicine, Stony Brook, New York
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Chattanooga Bariatrics, Chattanooga, Tennessee
  - Midsouth Bariatrics, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 711 subjects signed an informed consent form to participate in the study and proceeded to the screening eligibility process
Pre-assignment Details: 430 subjects randomized in a Treatment or Control group, 387 subjects received an Obalon Balloon or Sham Device.
Groups:
- Obalon Treatment Group: Obalon Balloon Device with Weight Loss Behavior Modification (WLBM) Program for 24 weeks
- Sham Control Group: Sham Device with Weight Loss Behavior Modification (WLBM) Program for 24 weeks
Period: Overall Study
Arm/Group | Obalon Treatment Group | Sham Control Group
Started (Subjects, Registered Dietitians and Adverse Event Assessors were blinded of device assignment) | 198 | 189
Completed Phase I (Week 24) (Device assignment unblinding and Obalon Balloon removal for Treatment Group) | 182 | 179
Crossover (Week 24) (Sham Group received Obalon Balloon & Treatment Group followed after balloon removal (WLBM for both)) | 170 | 138
Completed (Completed Phase II (Week 48), Obalon Balloon removal for Sham Group) | 160 | 128
Not Completed | 38 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obalon Treatment Group | Sham Control Group | Total
Number analyzed (Participants) | 198 | 189 | 387
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (9.6) | 42.5 (9.3) | 42.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 170 | 341
  Male | 27 | 19 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 24 | 39
  Not Hispanic or Latino | 183 | 165 | 348
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 29 | 50
  White | 165 | 155 | 320
  More than one race | 11 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.2 (2.7) | 35.5 (2.7) | 35.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Least-Square Mean Difference in % Total Body Loss (TBL) Between the Obalon Treatment and Sham Control Groups
Description: Statistical test to determine if the least-square mean difference between the Obalon Treatment and Sham Control groups is greater than the 2.1% TBL superiority margin
Time Frame: 24 Weeks
Population: Per Protocol cohort which includes subjects with at least 2 devices for at least 18 weeks
Measure: Least Squares Mean (Standard Error); unit: %TBL
Arm/Group | Obalon Treatment Group | Sham Control Group
Number analyzed (Participants) | 185 | 181
%TBL | 6.86 (0.37) | 3.59 (0.37)
Statistical Analysis 1: Comparison: Obalon Treatment Group vs Sham Control Group; Test type: Superiority; p = 0.0261, ANCOVA; Least-Square Mean Difference = 3.28, 95% CI 2-sided [2.24 to 4.32]

2. Primary Outcome: Percentage of Subjects in the Obalon Treatment Group With at Least 5% Total Body Loss (TBL)
Description: Statistical test to determine if the percentage of subjects in the Obalon Treatment and Sham Control with at least 5% Total Body Loss (TBL) is greater than 35%
Time Frame: 6 months
Population: Per Protocol cohort which includes subjects in the Obalon Treatment group with at least 2 balloons for at least 18 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Obalon Treatment Group: Subjects who received the Obalon Balloons.
Arm/Group | Obalon Treatment Group
Number analyzed (Participants) | 185
Participants | 120
Statistical Analysis 1: Comparison: Obalon Treatment Group; Subjects in the Obalon Treatment group with at least 2 Balloons and balloon therapy for at least 18 weeks; Test type: Superiority; p < 0.0001, Exact Test; Exact Confidence Interval = 64.9, 95% CI 2-sided [57.5 to 71.7]

3. Other Pre Specified Outcome: Percentage of Subjects With at Least 5% Total Body Loss: Obalon - Sham Group
Description: Difference in percentage of subjects between the Obalon Treatment and Sham Control groups with at least 5% Total Body Loss (TBL)
Time Frame: 6 Months
Population: Per Protocol cohort which includes subjects with at least 2 devices for at least 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Obalon Treatment Group | Sham Control Group
Number analyzed (Participants) | 185 | 181
Participants | 120 | 58
Statistical Analysis 1: Comparison: Obalon Treatment Group vs Sham Control Group; Test type: Superiority; p < 0.0001, Chi-squared; Percentage Difference = 32.8, 95% CI 2-sided [23.1 to 42.5]

ADVERSE EVENTS:
Time Frame: Six months
Groups:
- Treated Subjects: Treated subjects include the 198 subjects in Phase I of the study who received at least 1 Obalon Balloon and the 138 subjects in Phase II who crossover and received at least 1 Obalon Balloon
- Control Subjects: Control subjects include the 189 subjects in Phase I of the study who received at least 1 Sham Device and the 170 subjects in Phase II who were followed after balloon removal
Arm/Group | Treated Subjects | Control Subjects
All-Cause Mortality (participants affected / at risk) | 0/336 | 0/359
Serious Adverse Events (participants affected / at risk) | 7/336 | 5/359
Other Adverse Events (participants affected / at risk) | 321/336 | 221/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=336) | Control Subjects (N=359)
Peptic ulcer disease (Gastrointestinal disorders) | 1 (1) | 0 (0) — Device or Procedure Related
Abnormal Pap Smear (Reproductive system and breast disorders) | 1 (1) | 0 (0) — NOT Device or Procedure Related
Synovectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — NOT Device or Procedure Related
Breast Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) — NOT Device or Procedure Related
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) — NOT Device or Procedure Related
Bacterial Meningitis (Infections and infestations) | 1 (1) | 0 (0) — NOT Device or Procedure Related
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) — NOT Device or Procedure Related
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) — NOT Device or Procedure Related
Knee Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) — NOT Device or Procedure Related
Chiari Malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — NOT Device or Procedure Related
Heel Exostosis (General disorders) | 0 (0) | 1 (1) — NOT Device or Procedure Related
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — NOT Device or Procedure Related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=336) | Control Subjects (N=359)
Abdominal Pain (Gastrointestinal disorders) | 246 (501) | 51 (65) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 244/336 (76.62%) / 494 Events
Nausea (Gastrointestinal disorders) | 191 (315) | 37 (43) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 188/336 (55.95%) / 311 Events
Vomiting (Gastrointestinal disorders) | 61 (75) | 16 (16) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 58/336 (17.26%) / 71 Events
Dyspepsia (Gastrointestinal disorders) | 60 (73) | 10 (11) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 57/336 (16.96%) / 69 Events
Abdominal Distension (Gastrointestinal disorders) | 49 (54) | 10 (12) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 49/336 (14.58%) / 54 Events
Eructation (Gastrointestinal disorders) | 31 (37) | 0 (0) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 31/336 (9.23%) / 37 Events
Diarrhea (Gastrointestinal disorders) | 41 (47) | 15 (16) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 28/336 (8.33%) / 30 Events
Gastric Irritation (Gastrointestinal disorders) | 24 (25) | 0 (0) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 24/336 (7.14%) / 25 Events
Gastric Bleeding/Abrasion (Gastrointestinal disorders) | 17 (17) | 0 (0) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 17/336 (5.06%) / 17 Events
Constipation (Gastrointestinal disorders) | 51 (57) | 37 (47) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 9/336 (2.68%) / 10 Events
Common Cold/Upper Respiratory Infection (Infections and infestations) | 46 (56) | 44 (50) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 0/336 (0.00%) / 0 Events
Stomach/Seasonal Flu (Infections and infestations) | 29 (32) | 25 (28) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 0/336 (0.00%) / 0 Events
Headache/Migraine (Metabolism and nutrition disorders) | 22 (25) | 26 (30) — Treated Subjects - Device or Procedure Related Only (FDA Reviewed): 6/336 (1.79%) / 7 Events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes